CLINICAL TRIAL: NCT00092872
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety, Tolerability, and Efficacy of MK0557 in Obese Patients
Brief Title: A 1-Year Study of an Investigational Drug in Obese Patients (0557-012)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0557-012; MK0557-012; 2004_031
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — spiro(cyclohexane-1,3'(1'H)-furo(3,4-C)pyridine)-4-carboxamide, N-(1-(2-fluorophenyl)-1h-pyrazol-3-yl)-1'-oxo-, trans-

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0557

SUMMARY:
This is a 1-year study to assess the safety, tolerability, and efficacy of an investigational drug in obese patients after a very low calorie diet.

ELIGIBILITY:
Inclusion Criteria:

* Obese men and nonpregnant women between the ages of 18 and 65 years with a body mass index (height to weight ratio) as required by the study.

Exclusion Criteria:

* Patients with uncontrolled high blood pressure and/or diabetes mellitus (high blood sugar)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2003-11; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Body weight after 1 year of treatment. | After 1 year of treatment
Safety and tolerability. | After 1 year of treatment

SECONDARY OUTCOMES:
Waist circumference; Blood pressure, body fat mass, biochemical markers (fasting plasma, lipid profile, fasting plasma glucose, leptin, insulin, insulin sensitivity); body weight after 2 years | After 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Erondu N, Gantz I, Musser B, Suryawanshi S, Mallick M, Addy C, Cote J, Bray G, Fujioka K, Bays H, Hollander P, Sanabria-Bohorquez SM, Eng W, Langstrom B, Hargreaves RJ, Burns HD, Kanatani A, Fukami T, MacNeil DJ, Gottesdiener KM, Amatruda JM, Kaufman KD, Heymsfield SB. Neuropeptide Y5 receptor antagonism does not induce clinically meaningful weight loss in overweight and obese adults. Cell Metab. 2006 Oct;4(4):275-82. doi: 10.1016/j.cmet.2006.08.002. PMID 17011500